CLINICAL TRIAL: NCT05363150
Title: Feasibility of a Smart Device Application for Home-based Prehabilitation in Patients Undergoing Lung Cancer Surgery: A Prospective Observational Pilot Study
Brief Title: Feasibility of a Smart Device Application for Home-based Prehabilitation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Susie Yoon, Professor, Seoul National University Hospital
Other Study IDs: Prehab_app
Record Dates: First submitted 2022-05-03; First posted 2022-05-05 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Cancer; Prehabilitation
Keywords: Cancer patient; Cancer Surgery; Prehabilitation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the feasibility of a home-based exercise training program using a smartphone application in patients planning for cancer surgery, and to determine the effectiveness of this application on functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (19-70) who are scheduled for elective cancer surgery
* American Society of Anesthesiologists (ASA) physical status classification I or II
* Patients who can use a smartphone application
* Patients who can perform an exercise program for at least 3 weeks from the first visit to the preoperative clinic to elective surgery

Exclusion Criteria:

* Patients who are unable to communicate
* Patients under the age of 19 and over 70
* Patients who have a major medical or psychiatric disorder that is expected to affect exercise
* Patients with contraindications to the general rehabilitation program

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visits preoperative evaluation clinic for preoperative counseling before the cancer surgery
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Compliance of a smartphone application | A day before surgery at ward
  Based on the data saved in the application, when the program started and ended, how many steps and distance the patient exercised per day, how many sets patient did muscle exercise per day and week will be collected to calculate the compliance.
Satisfaction of a smartphone application | A day before surgery at ward
  Using the questionnaire that we made to evaluation the satisfaction of a smartphone application.

SECONDARY OUTCOMES:
Korean-EORTC QLQ C-30 | 4 weeks before the surgery at clinic, a day before the surgery at ward
  EORTC QLQ C-30: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaires Core-30
  A questionnaire which is designed to assess the different aspects that define the QoL of cancer patients. (Total score ranging 0 to 100, A high score for a functional scale represents a high level of functioning)
6-minute walk test | 4 weeks before the surgery at clinic, a day before the surgery at ward
  The distance that patient can walk during 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Susie Yoon, PhD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided